CLINICAL TRIAL: NCT01890070
Title: Study of the Nutraceutical Properties and Health Benefits of Traditional Components of the Mediterranean Diet - A Cross Over Interventional Study
Brief Title: Study of the Nutraceutical Properties and Health Benefits of Traditional Components of the Mediterranean Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, LAURA DI RENZO, Professor of Human Nutrition, University of Rome Tor Vergata
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DM 06/12/2011 n° prot. 32064
Record Dates: First submitted 2013-06-24; First posted 2013-07-01 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Obesity
Keywords: mediterranean diet, nutrigenomics, body composition, inflammation, oxidative stress
MeSH Terms: conditions — Obesity; Inflammation | interventions — Chocolate; whole grape extract; Olive Oil; horse chestnut seed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (28):
- STANDARD DIET (Placebo Comparator): each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  Standard diet (Mediterrean reference: carbohydrates 55%-60%; protein 15% - 20% of which 50% are of vegetable derivation; total fats < 30% e 30 g of fiber)
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Other: No Dietary Supplement
- STANDARD DIET WITH HAZELNUTS (Experimental): Intervention type: each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  Standard diet (Mediterrean reference: carbohydrates 55%-60%; protein 15% - 20% of which 50% are of vegetable derivation; total fats < 30% e 30 g of fibers) with 40g Italian hazelnuts from Piedmont with Protected Geographical Indication Certification
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Hazelnuts
- STANDARD DIET WITH RED WINE (Experimental): Intervention type: each patient is administered a food plan for four weeks. Every patient is required to consume per day :
  Standard diet (Mediterrean reference: carbohydrates 55%-60%; protein 15% - 20% of which 50% are of vegetable derivation; total fats < 30% e 30 g of fibers) with 200 ml of Italian organic Red Wine.
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Red wine
- STANDARD DIET WITH CHESTNUTS (Experimental): Intervention type: each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  Standard diet (Mediterrean reference: carbohydrates 55%-60%; protein 15% - 20% of which 50% are of vegetable derivation; total fats < 30% e 30 g of fibers) with 100 g of Italian organic chestnuts.
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Chestnut
- STANDARD DIET WITH CHOCOLATE (Experimental): Intervention type: each patient is administered a food plan for four weeks. Every patient is required to consume per day :
  Standard diet (Mediterrean reference: carbohydrates 55%-60%; protein 15% - 20% of which 50% are of vegetable derivation; total fats < 30% e 30 g of fibers) with 100 g of Extra-dark Italian Chocolate (min. 70% of organic cocoa solids)
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Chocolate
- STANDARD DIET WITH WILD MIXED GREEN (Experimental): Intervention type: each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  Standard diet (Mediterrean reference: carbohydrates 55%-60%; protein 15% - 20% of which 50% are of vegetable derivation; total fats < 30% e 30 g of fibers) with 200 g of Italian organic wild mixed green
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Wild mixed greens
- STANDARD DIET WITH OLIVE OIL (Experimental): Intervention type: each patient is administered a food plan for four weeks. Every patient patient is required to consume per day :
  Standard diet (Mediterrean reference: carbohydrates 55%-60%; protein 15% - 20% of which 50% are of vegetable derivation; total fats < 30% e 30 g of fibers) with 100g of Italian organic Olive Oil
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Olive Oil
- HIGH FAT DIET (Placebo Comparator): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High fat diet (carbohydrates 35%; protein 15%; total fats 50%)
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Other: No Dietary Supplement
- HIGH FAT WITH HAZELNUTS (Experimental): Intervention type: each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High fat diet (carbohydrates 35%; protein 15%; total fats 50%) with 40g of Italian hazelnuts from Piedmont with Protected Geographical Indication Certification.
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Hazelnuts
- HIGH FAT WITH RED WINE (Experimental): Intervention type: each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High fat diet (carbohydrates 35%; protein 15%; total fats 50%)with 200 ml of Italian organic Red Wine
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Red wine
- HIGH FAT WITH CHESTNUT (Experimental): Intervention type: each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High fat diet (carbohydrates 35%; protein 15%; total fats 50%) with 100 g of Italian organic chestnuts.
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Chestnut
- HIGH FAT WITH CHOCOLATE (Experimental): Intervention type: each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High fat diet (carbohydrates 35%; protein 15%; total fats 50%) with 100 g of Extra-dark Italian Chocolate (min. 70% of organic cocoa solids)
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Chocolate
- HIGH FAT WITH WILD MIXED GREEN (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High fat diet (carbohydrates 35%; protein 15%; total fats 50%) with 200 g of Italian organic wild mixed green
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Wild mixed greens
- HIGH FAT WITH OLIVE OIL (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High fat diet (carbohydrates 35%; protein 15%; total fats 50%) with 100 of Italian organic Olive oil
  Three weeks of washout to avoid additive effects on treatment following.
  Interventions: Dietary Supplement: Olive Oil
- LOW CARBOHYDRATE DIET (Placebo Comparator): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  Low carbohydrate diet (carbohydrates 35%; protein 30%; total fats 35%)
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Other: No Dietary Supplement
- LOW CARBOHYDRATE DIET WITH HAZELNUT (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  Low carbohydrate diet (carbohydrates 35%; protein 30%; total fats 35%) with 40g Italian hazelnuts from Piedmont with Protected Geographical Indication Certification
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Hazelnuts
- LOW CARBOHYDRATE DIET WITH RED WINE (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  Low carbohydrate diet (carbohydrates 35%; protein 30%; total fats 35%) with 200 ml of Italian organic Red Wine
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Red wine
- LOW CARBOHYDRATE DIET WITH CHESTNUT (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  Low carbohydrate diet (carbohydrates 35%; protein 30%; total fats 35%) with 100 g of Italian organic chestnuts
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Chestnut
- LOW CARBOHYDRATE DIET CHOCOLATE (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  Low carbohydrate diet (carbohydrates 35%; protein 30%; total fats 35%) with 100 g of Extra-dark Italian Chocolate (min. 70% of organic cocoa solids)
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Chocolate
- LOW CARBOHYDRATE DIET WITH WILD MIXED GREEN (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  Low carbohydrate diet (carbohydrates 35%; protein 30%; total fats 35%) with 200 g of Italian organic wild mixed green
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Wild mixed greens
- LOW CARBOHYDRATE DIET WITH OLIVE OIL (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  Low carbohydrate diet (carbohydrates 35%; protein 30%; total fats 35%) with 100 of Italian organic Olive Oil
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Olive Oil
- HIGH PROTEIN DIET (Placebo Comparator): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High protein diet (carbohydrates 30%; protein 40%; total fats 30%)
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Other: No Dietary Supplement
- HIGH PROTEIN DIET WITH HAZELNUT (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High protein diet (carbohydrates 30%; protein 40%; total fats 30%) with 40g Italian hazelnuts from Piedmont with Protected Geographical Indication Certification
  Interventions: Dietary Supplement: Hazelnuts
- HIGH PROTEIN DIET WITH RED WINE (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High protein diet (carbohydrates 30%; protein 40%; total fats 30%) with 200 ml of Italian organic Red Wine
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Red wine
- HIGH PROTEIN DIET WITH CHESTNUT (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High protein diet (carbohydrates 30%; protein 40%; total fats 30%) with 100 g of Italian organic chestnuts
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Chestnut
- HIGH PROTEIN DIET WITH CHOCOLATE (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High protein diet (carbohydrates 30%; protein 40%; total fats 30%) with 100 g of Extra-dark Italian Chocolate (min. 70% of organic cocoa solids)
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Chocolate
- HIGH PROTEIN DIET WITH ITALIAN ORGANIC WILD MIXED GREEN (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High protein diet (carbohydrates 30%; protein 40%; total fats 30%) with 200 g of Italian organic wild mixed green
  Three weeks of washout to avoid additive effects on treatments to follow.
  Interventions: Dietary Supplement: Wild mixed greens
- HIGH PROTEIN DIET WITH OLIVE OIL (Experimental): Intervention type: Each patient is administered a food plan for four weeks. Every patient is required to consume per day:
  High protein diet (carbohydrates 30%; protein 40%; total fats 30%) with 100 of Italian organic Olive Oil
  This is followed by a 3 week wash out period, to neutralize any additive effects.
  Interventions: Dietary Supplement: Olive Oil

INTERVENTIONS:
Dietary Supplement: Hazelnuts — Italian hazelnuts from Piedmont with Protected Geographical Indication Certification
  Other Names: Corylus avellana
  Arms: HIGH FAT WITH HAZELNUTS; HIGH PROTEIN DIET WITH HAZELNUT; LOW CARBOHYDRATE DIET WITH HAZELNUT; STANDARD DIET WITH HAZELNUTS
Dietary Supplement: Chocolate — Extra-dark Italian Chocolate (min. 70% of organic cocoa solids)
  Other Names: Theobroma cacao
  Arms: HIGH FAT WITH CHOCOLATE; HIGH PROTEIN DIET WITH CHOCOLATE; LOW CARBOHYDRATE DIET CHOCOLATE; STANDARD DIET WITH CHOCOLATE
Dietary Supplement: Red wine — Italian Organic Red Wine
  Other Names: Vitis vinifera
  Arms: HIGH FAT WITH RED WINE; HIGH PROTEIN DIET WITH RED WINE; LOW CARBOHYDRATE DIET WITH RED WINE; STANDARD DIET WITH RED WINE
Dietary Supplement: Olive Oil — Italian Organic Olive Oil
  Other Names: Olea europea
  Arms: HIGH FAT WITH OLIVE OIL; HIGH PROTEIN DIET WITH OLIVE OIL; LOW CARBOHYDRATE DIET WITH OLIVE OIL; STANDARD DIET WITH OLIVE OIL
Dietary Supplement: Wild mixed greens — Italian organic wild mixed greens
  Other Names: Chicory, rocket, nettle
  Arms: HIGH FAT WITH WILD MIXED GREEN; HIGH PROTEIN DIET WITH ITALIAN ORGANIC WILD MIXED GREEN; LOW CARBOHYDRATE DIET WITH WILD MIXED GREEN; STANDARD DIET WITH WILD MIXED GREEN
Dietary Supplement: Chestnut — Italian Organic Chestnut
  Other Names: Castanea sativa
  Arms: HIGH FAT WITH CHESTNUT; HIGH PROTEIN DIET WITH CHESTNUT; LOW CARBOHYDRATE DIET WITH CHESTNUT; STANDARD DIET WITH CHESTNUTS
Other: No Dietary Supplement — Mediterranean Reference Diet, High Fat Diet, Low Carbohydrate or High Protein Diet without an added dietary supplement (hazelnut, chocolate, red wine, wild mixed greens, chestnuts, olive oil)
  Arms: HIGH FAT DIET; HIGH PROTEIN DIET; LOW CARBOHYDRATE DIET; STANDARD DIET

SUMMARY:
The present protocol is designed to conduct nutrigenomic and nutrigenetic studies on foods conforming to the Mediterranean diet, in order to determine the effect functional foods have on blood parameters (cholesterol metabolism, glucose metabolism, hepatic function, inflammation, nutritional status) and body composition in the context of four different diets (standard, high fat, high protein, low carbohydrate). The study focuses on the effect of these nutraceutical foods in relation to different diets. Diets were chosen to reflect the standard reference diets used by the general population, so as the outcomes of the addition of each interventional food element may be interpreted in the context of a variety of dietary patterns.

DETAILED DESCRIPTION:
This study envisages the enrollment of subjects, to be recruited consecutively from May 2013 to May 2015 from the staff of the laboratory of the Evaluation of Nutritional State, Nutrigenetics and nutrigenomics of the Human Nutrition and Diet section of the University of Rome Tor Vergata.

The study will be conducted in accordance with the Declaration of Helsinki, and approved by the Committee of the Ministero delle Politiche Alimentari e Forestali (MIPAAF) , Italy, approved by DM 06/12/2011 n° prot. 32064. All participants will be required to provide written informed consent for the study.

At the time of recruitment, relevant subject data will be collected including clinical history, dietary habits, pharmacological therapy, smoking habit, alcohol consumption and level of physical activity.

Exclusion criteria include history of coronary vascular disease, peripheral or cerebro- vascular disease, hepatic disease, diagnosis of diabetes mellitus, autoimmune disease, immunodeficiency syndrome or malignant neoplasia.

The subjects enrolled will undergo:

* Anthropometric measures (body weight, height, waist, hip, abdominal, neck, arm and forearm circumferences).
* Skin fold measurements (bicipital, tricipital, subscapular, pectoral, supra iliac, abdominal, anterior thigh, internal thigh, supra patellar and popliteal);
* Blood Pressure;
* Body composition evaluation (bone, fat and lean mass), evaluated by DEXA (iDXA; GE
* Medical Systems, Milwaukee, WI) (Dual energy X-ray Absorptiometry; DPX Lunar Radiation Corp., Madison, Wisconsin, USA);
* Distribution of body fluids, evaluated by bioimpedensometry. Resistance, reactance, phase angle at 50 kHz will be measured using the Bioelectrical Impedance Analysis method (BIA 101S, by Akern/RIL System-Florence
* Analysis of genetic expression Participants will be randomized into groups.

Each group will cycle through different interventions, according to a cross over study. The interventions are represented by different dietary plans based on different meals, consisting of:

1. Standard Diet (SD) alone, and SD with functional food (40g of hazelnuts or 150 ml of biological red wine, or 100g of chestnuts, or 200g of wild mixed greens, or 100 g of olive oil, or 100 g of chocolate);
2. High Fat diet (HF) alone, and HF with functional food (40g of hazelnuts or 150 ml of biological red wine, or 100g of chestnuts, or 200g of wild mixed greens, or 100 g of olive oil, or 100 g of chocolate).
3. Low Carbohydrate diet (LC) alone, and LC with functional food (40g of hazelnuts or 150 ml of biological red wine, or 100g of chestnuts, or 200g of wild mixed greens, or 100 g of olive oil, or 100 g of chocolate).
4. High Protein (HP) alone, and HP with functional food (40g of hazelnuts or 150 ml of biological red wine, or 100g of chestnuts, or 200g of wild mixed greens, or 100 g of olive oil, or 100 g of chocolate).

The duration of the experimental period is 4 weeks for each diet, with a wash-out period of 3 weeks at the beginning of the study between one diet and the next.

ELIGIBILITY:
Inclusion Criteria:Age:

18 to 75 years inclusive BMI >19 kg/m2

-

Exclusion Criteria:

* Past history of ischaemic coronary artery disease
* Peripheral or cerebral vasculopathy
* Hepatic disease
* Diabetes Mellitus
* Autoimmune disease
* HIV/AIDS
* Neoplastic disease
* Use of the following medications: lipid-lowering medications, oral anti-diabetic medication or insulin, nitroglycerin, corticosteroids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Sarcopenic index | Variation in sarcopenic index from baseline to 4 weeks
  To calculate the sarcopenic index three calculations will be made: Body Cell Mass Index from bioelectrical impedance analysis (body cell mass in kilograms divided by height in metres squared),and the Appendicular Skeletal Muscle Index (sum of appendicular muscle mass divided by height in metres squared)and Relative Skeletal Muscle Index (total body lean mass divided by height in metres squared)both calculated from dual-energy X-ray asorptiometry.

SECONDARY OUTCOMES:
Cardiovascular Risk Index | Variation in cardiovascular risk index from baseline to 4 weeks
  Cardiovascular Risk Index will be calculated from 3 formulas: Total Cholesterol (mg/dl) divided by High Density Lipoprotein (mg/dl), Low Density Lipoprotein (mg/dl) divided by High Density Lipoprotein (mg/dl), Log10 Triglycerides (mg/dl) divided by High Density Lipoprotein (mg/dl)
Homeostatic Model Assessment (HOMA-IR) | Variation in HOMA from baseline to 4 weeks
  HOMA will be calculated as follows: Blood glucose (mmol/L) x Blood Insulin (mU/L) divided by 22.5
Prognostic Inflammatory and Nutritional Index (PINI) | Variation in PINI from baseline to 4 weeks
  PINI will be calculated as follows: [C-reactive Protein (mg/L) multiplied by alpha-1 acid glycoprotein (g/L)] divided by [albumin (g/L) multiplied by prealbumin (g/L)]
Nuclear factor kappa-light-chain-enhancer of activated B cells (NFkappaB) | Variation in expression of NFkappaB from baseline to 4 weeks
  Measurement of gene up-regulation or down-regulation in order of magnitude set at ±2FC (fundamental-costant-based system of units)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition and Nutrigenomic, School of Medicine University of Rome Torvergata, Rome, Rome, Italy

REFERENCES:
- [Derived] Di Renzo L, Frank G, Pala B, Cianci R, De Santis GL, Nicoletti F, Bigioni G, Ortoman M, Borro M, Simmaco M, Peluso D, De Lorenzo A, Gualtieri P. Characterization of Gut Microbiota Profile in Lipedema: A Pilot Study. Nutrients. 2025 Dec 13;17(24):3909. doi: 10.3390/nu17243909. PMID 41470854
- [Derived] Di Renzo L, Gualtieri P, Frank G, Cianci R, Raffaelli G, Peluso D, Bigioni G, De Lorenzo A. Sex-Specific Adherence to the Mediterranean Diet in Obese Individuals. Nutrients. 2024 Sep 12;16(18):3076. doi: 10.3390/nu16183076. PMID 39339676
- [Derived] Gualtieri P, Marchetti M, Frank G, Smeriglio A, Trombetta D, Colica C, Cianci R, De Lorenzo A, Di Renzo L. Antioxidant-Enriched Diet on Oxidative Stress and Inflammation Gene Expression: A Randomized Controlled Trial. Genes (Basel). 2023 Jan 13;14(1):206. doi: 10.3390/genes14010206. PMID 36672947
- [Derived] Marchetti M, Gualtieri P, De Lorenzo A, Trombetta D, Smeriglio A, Ingegneri M, Cianci R, Frank G, Schifano G, Bigioni G, Di Renzo L. Dietary omega-3 intake for the treatment of morning headache: A randomized controlled trial. Front Neurol. 2022 Sep 20;13:987958. doi: 10.3389/fneur.2022.987958. eCollection 2022. PMID 36203988
- [Derived] Perrone MA, Gualtieri P, Gratteri S, Ali W, Sergi D, Muscoli S, Cammarano A, Bernardini S, Di Renzo L, Romeo F. Effects of postprandial hydroxytyrosol and derivates on oxidation of LDL, cardiometabolic state and gene expression: a nutrigenomic approach for cardiovascular prevention. J Cardiovasc Med (Hagerstown). 2019 Jul;20(7):419-426. doi: 10.2459/JCM.0000000000000816. PMID 31593559
- [Derived] Di Renzo L, Cioccoloni G, Falco S, Abenavoli L, Moia A, Sinibaldi Salimei P, De Lorenzo A. Influence of FTO rs9939609 and Mediterranean diet on body composition and weight loss: a randomized clinical trial. J Transl Med. 2018 Nov 12;16(1):308. doi: 10.1186/s12967-018-1680-7. PMID 30419927
- [Derived] Colica C, Avolio E, Bollero P, Costa de Miranda R, Ferraro S, Sinibaldi Salimei P, De Lorenzo A, Di Renzo L. Evidences of a New Psychobiotic Formulation on Body Composition and Anxiety. Mediators Inflamm. 2017;2017:5650627. doi: 10.1155/2017/5650627. Epub 2017 Sep 24. PMID 29147070
- [Derived] Colica C, Di Renzo L, Trombetta D, Smeriglio A, Bernardini S, Cioccoloni G, Costa de Miranda R, Gualtieri P, Sinibaldi Salimei P, De Lorenzo A. Antioxidant Effects of a Hydroxytyrosol-Based Pharmaceutical Formulation on Body Composition, Metabolic State, and Gene Expression: A Randomized Double-Blinded, Placebo-Controlled Crossover Trial. Oxid Med Cell Longev. 2017;2017:2473495. doi: 10.1155/2017/2473495. Epub 2017 Aug 9. PMID 28855976
- [Derived] De Lorenzo A, Costacurta M, Merra G, Gualtieri P, Cioccoloni G, Marchetti M, Varvaras D, Docimo R, Di Renzo L. Can psychobiotics intake modulate psychological profile and body composition of women affected by normal weight obese syndrome and obesity? A double blind randomized clinical trial. J Transl Med. 2017 Jun 10;15(1):135. doi: 10.1186/s12967-017-1236-2. PMID 28601084
- [Derived] Colica C, Merra G, Gasbarrini A, De Lorenzo A, Cioccoloni G, Gualtieri P, Perrone MA, Bernardini S, Bernardo V, Di Renzo L, Marchetti M. Efficacy and safety of very-low-calorie ketogenic diet: a double blind randomized crossover study. Eur Rev Med Pharmacol Sci. 2017 May;21(9):2274-2289. PMID 28537652
- [Derived] Di Renzo L, Merra G, Botta R, Gualtieri P, Manzo A, Perrone MA, Mazza M, Cascapera S, De Lorenzo A. Post-prandial effects of hazelnut-enriched high fat meal on LDL oxidative status, oxidative and inflammatory gene expression of healthy subjects: a randomized trial. Eur Rev Med Pharmacol Sci. 2017 Apr;21(7):1610-1626. PMID 28429343
- [Derived] De Lorenzo A, Bernardini S, Gualtieri P, Cabibbo A, Perrone MA, Giambini I, Di Renzo L. Mediterranean meal versus Western meal effects on postprandial ox-LDL, oxidative and inflammatory gene expression in healthy subjects: a randomized controlled trial for nutrigenomic approach in cardiometabolic risk. Acta Diabetol. 2017 Feb;54(2):141-149. doi: 10.1007/s00592-016-0917-2. Epub 2016 Oct 5. PMID 27709360
- [Derived] Di Renzo L, Tyndall E, Gualtieri P, Carboni C, Valente R, Ciani AS, Tonini MG, De Lorenzo A. Association of body composition and eating behavior in the normal weight obese syndrome. Eat Weight Disord. 2016 Mar;21(1):99-106. doi: 10.1007/s40519-015-0215-y. Epub 2015 Sep 7. PMID 26347355
- [Derived] Di Renzo L, Marsella LT, Sarlo F, Soldati L, Gratteri S, Abenavoli L, De Lorenzo A. C677T gene polymorphism of MTHFR and metabolic syndrome: response to dietary intervention. J Transl Med. 2014 Nov 29;12:329. doi: 10.1186/s12967-014-0329-4. PMID 25432492
- [Derived] Di Renzo L, Carraro A, Valente R, Iacopino L, Colica C, De Lorenzo A. Intake of red wine in different meals modulates oxidized LDL level, oxidative and inflammatory gene expression in healthy people: a randomized crossover trial. Oxid Med Cell Longev. 2014;2014:681318. doi: 10.1155/2014/681318. Epub 2014 Apr 30. PMID 24876915